CLINICAL TRIAL: NCT01127035
Title: STUDIO IN DOPPIO CIECO DISODIOCROMOGLICATO + PLACEBO vs DISODIOCROMOGLICATO + IMMUNOTERAPIA SPECIFICA SUBLINGUALE PER ALTERNARIA IN PAZIENTI CON RINITE ALLERGICA DOVUTA A SENSIBILIZZAZIONE AD ALTERNARIA
Brief Title: Sublingual Immunotherapy In Alternaria-Induced Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Genova (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLITALT2004
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2008-01

CONDITIONS: Allergic Rhinitis (w/w Asthma) Due to Alternaria Alternata
Keywords: allergic rhinitis; alternaria alternata; symptom score
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Sublingual Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SLIT (Experimental): sublingual immunotherapy biologically standardized
  Interventions: Biological: sublingual immunotherapy
- placebo (Placebo Comparator): same preparation of SLIT without the allergen
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: sublingual immunotherapy
  Arms: SLIT
Biological: placebo
  Arms: placebo

SUMMARY:
Respiratory allergy due to Alternaria is a relevant clinical problem, and specific immunotherapy may represent a viable treatment option. Sublingual immunotherapy (SLIT) is safe and effective, but data for Alternaria are lacking. The study is aimed at assessing the efficacy of a standardized SLIT in patients sensitised to Alternaria, in a randomized, double blind, placebo controlled fashion.

Patients with rhinitis with/without intermittent asthma, and ascertained allergy to Alternaria are enrolled. After a baseline season, SLIT or matched placebo are given for 10 months. Symptoms and rescue medication intake are recorded on diary cards from June to October. Skin prick test, specific IgE and IgG4 and precipitins are measured at baseline and at the end of the study. Alternaria spore count is also performed. Primary outcome is the change in symptom score in the active vs placebo group. Secondary outcomes: changes in rescue medication intake, alternaria specific IgE and IgG4, skin prick test reactivity.

ELIGIBILITY:
Inclusion Criteria:

* Allergic rhinitis
* Symptoms May-October
* Specific IgE to alternaria (skin test/radioallergosorbent [RAST] test)
* Age >14

Exclusion Criteria:

* Sensitization to mites, parietaria, mugwort
* Pregnancy-lactation
* Malignancies
* Chronic systemic steroids
* Previous immunotherapy to alternaria

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
change in symptom score active versus placebo

SECONDARY OUTCOMES:
change in rescue medication intake

CONTACTS AND LOCATIONS:
Locations (1):
- Rimini Hospital, Rimini, Italy

REFERENCES:
- [Background] Tabar AI, Lizaso MT, Garcia BE, Gomez B, Echechipia S, Aldunate MT, Madariaga B, Martinez A. Double-blind, placebo-controlled study of Alternaria alternata immunotherapy: clinical efficacy and safety. Pediatr Allergy Immunol. 2008 Feb;19(1):67-75. doi: 10.1111/j.1399-3038.2007.00589.x. Epub 2007 Jul 25. PMID 17651380
- [Derived] Cortellini G, Spadolini I, Patella V, Fabbri E, Santucci A, Severino M, Corvetta A, Canonica GW, Passalacqua G. Sublingual immunotherapy for Alternaria-induced allergic rhinitis: a randomized placebo-controlled trial. Ann Allergy Asthma Immunol. 2010 Nov;105(5):382-6. doi: 10.1016/j.anai.2010.08.007. Epub 2010 Sep 26. PMID 21055665